CLINICAL TRIAL: NCT04857463
Title: The Effects of Continuous Intake of ONS on the Nutritional Status of Taiwanese Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Meiji Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: N202011065
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-01

CONDITIONS: Malnutrition Elderly
Keywords: Sarcopenia, Oral nutritional supplement, elderly people, nutritional education, malnutrition risk
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: This study was a clustered, randomized, parallel, multicenter clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nutritional supplement drink (Experimental): Nutritional supplement, this group receives a nutritional supplement for a period of 12 weeks.
  Interventions: Other: Nutritional supplement drink
- Nutritional education (Placebo Comparator): Qualified clinical dietitians provide regular nutrition education and ensure the effectiveness of nutrition education
  Interventions: Other: Nutritional education
- Healthy control (No Intervention): No intervention was done to this group, only blood collection, physical performance and anthropometric assessment were done.

INTERVENTIONS:
Other: Nutritional supplement drink — At the intervention period (0th to 12th week of the experiment), In addition to nutrition and health education, subjects were provided with 2 bottles of commercially available oral nutritional supplements (Meiji Mei Balance, Meiji Co., Ltd., Tokyo, Japan) every day, between lunch and dinner and before bedtime.
  Arms: Nutritional supplement drink
Other: Nutritional education — At the intervention period (0th to 12th week of the experiment) , subjects will be given regular nutrition education by a qualified clinical dietitian to ensure the effectiveness of nutrition education, in order for the nutrition education group to benefit from participating in this trial, the subjects will also be provided with the same nutritional products after the trial
  Arms: Nutritional education

SUMMARY:
Past studies have pointed out that adequate intake of calories and protein in the elderly can deferred sarcopenia and debilitating conditions. Therefore, this study intends to use oral nutrition as a way of nutritional supplements, without affecting the subjects' normal meal intake, and supplements with snacks It is expected that there will be benefits in protein and muscle synthesis.

However, the palatability of oral nutritional products will affect the effectiveness of nutritional supplements. Therefore, this test provides nutrients that are easy for the subjects to ingest with a variety of flavors, in order to achieve the test calories and protein needs.

In order to investigate and compare the nutritional status, serum zinc and vitamin D status in healthy (MUST score 0) elderly and at risk of malnutrition elderly, we recruited healthy elderlies in the nursing home.

DETAILED DESCRIPTION:
In this study, subjects were randomly assigned. Through a multi-center research method, a total of 100 eligible subjects were recruited, and their consent was obtained and a subject consent form was signed. The subjects were divided into two groups according to the way of nutritional intervention, including nutritional education (NE) and nutritional supplement drink (NSD), with 50 people in each group. The NE group is given regular nutrition education by qualified clinical nutritionists to ensure the effectiveness of nutrition education. In the NSD group, in addition to nutrition and health education, daily oral supplements (Meiji Mei Balance, Meiji Co., Ltd., Tokyo, Japan) are provided daily, and snacks are supplemented between lunch and dinner and before bedtime, 2 per day. bottle. The two groups were divided into groups by lottery, and the intervention period was 12 weeks. During the intervention period, blood will be drawn at the beginning, 6th, and 12th week of the case, and blood pressure, body position, body composition and muscle strength will be measured, and dietary intake will be assessed. At the same time, a quality of life survey will also be conducted. survey, QoL survey.

Moreover, we recruited 50 healthy elderly to investigate and compare the nutritional status, serum zinc and vitamin D status in healthy elderly and at risk of malnutrition elderly. This group was considered as a control group and we didn't do any intervention after blood collection and physical measurements.

ELIGIBILITY:
Inclusion Criteria:

1. age >65 years old (regardless of gender)
2. Malnutrition risk judgment: Subjects were assessed as moderate and high malnutrition risk with the malnutrition risk screening tool MUST (Malnutrition Universal Screening Tool)

Exclusion Criteria:

1. chronic diseases such as diabetes, end stage of chronic kidney disease, cancer.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 161 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Blood biochemical value | at the start of the experiment and at the 6th and 12th week
  blood cell analysis, liver function test (AST/ALT), blood sugar, triglycerides, nutritional indicators (serum albumin), kidney function (urea nitrogen, creatinine), vitamin D, zinc, etc
Blood pressure | at the start of the experiment and at the 6th and 12th week
  measure systolic and diastolic blood pressure.
Body position measurement | at the start of the experiment and at the 6th and 12th week
  height, weight, waist-to-hip ratio, body mass index, etc.
Body composition | at the start of the experiment and at the 6th and 12th week
  Use a body fat machine to measure muscle mass, fat mass and water content.
Muscle strength test | at the start of the experiment and at the 6th and 12th week
  measure 6m walking speed, grip strength measurement, etc.
Diet pattern | at the start of the experiment and at the 6th and 12th week
  Evaluate the 24-hour recall method and Three-day dietary record
Quality of life and health status | at the start of the experiment and at the 6th and 12th week
  Use the quality of life questionnaire (SF-36) to evaluate the quality of life and health status

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan